CLINICAL TRIAL: NCT00848562
Title: Oral Nicorandil to Reduce Cardiac Death After Coronary Revascularization in Hemodialysis Patients: A Randomized Trial
Brief Title: Nicorandil Study to Reduce Cardiac Death After Percutaneous Coronary Intervention (PCI) in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toujinkai Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NICO-HDPCI-1
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Acute Myocardial Infarction; Congestive Heart Failure
Keywords: sudden cardiac death
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac | interventions — Nicorandil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nicorandil (Experimental)
  Interventions: Drug: Nicorandil

INTERVENTIONS:
Drug: Nicorandil — Oral administration of nicorandil (15 mg/day)

SUMMARY:
Survival after invasive coronary revascularization is worse in patients with chronic kidney disease than in those without it. The investigators aimed to examine whether oral administration of nicorandil, a hybrid of nitrate and adenosine triphosphate-sensitive potassium channel opener, could improve the survival of end-stage renal disease patients with coronary artery disease by inhibiting cardiac death after coronary revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients with coronary artery disease who had undergone a successful first PCI with bare-metal stents between July 1, 2001 and December 31, 2003.

Exclusion Criteria:

* Subjects with moderate or worse cardiac valvular disease or old myocardial infarction at the point of first PCI.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2002-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Cardiac death (sudden cardiac death, deaths due to acute myocardial infarction or congestive heart failure) | Jan 1, 2002 to Dec 31, 2006

SECONDARY OUTCOMES:
All-cause mortality | Jan 1, 2002 to Dec 31, 2006

CONTACTS AND LOCATIONS:
Locations (1):
- Toujinkai Hospital, Kyoto, Kyoto, Japan